CLINICAL TRIAL: NCT00862719
Title: A Phase II Trial of Inhibition of CD26 Peptidase Using Sitagliptin to Enhance Engraftment After Umbilical Cord Blood Transplantation for Adults With Hematological Malignancies
Brief Title: Sitagliptin Umbilical Cord Blood Transplant Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0812-15; IUCRO-0223
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Results first posted 2016-08-04 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Leukemia, Myeloid, Acute; Acute Lymphoblastic Leukemia; Myelodysplasia; Leukemia, Myelogenous, Chronic; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sitagliptin once per day (Experimental): 600 mg sitagliptin once per day orally starting on Day -1 for a total of 4 doses
  Interventions: Drug: Sitagliptin
- Sitagliptin twice per day (Experimental): 600 mg sitagliptin twice per day orally starting on Day -1 for a total of 8 doses
  Interventions: Drug: Sitagliptin
- Sitagliptin three times per day (Experimental): 600 mg sitagliptin three times per day orally starting on Day -1 for a total of 12 doses
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — 600 mg sitagliptin taken orally per the schedule listed in each of the three separate arms.
  Other Names: Januvia

SUMMARY:
The main purpose of this trial is to study whether the drug sitagliptin can be given safely to patients undergoing umbilical cord blood transplantation to speed up engraftment (recovery of blood counts after transplant).

DETAILED DESCRIPTION:
Umbilical cord blood (UCB) is increasingly used as a source of stem cells for patients with blood cancers who need an allogeneic stem cell transplant (a transplant with stem cells from another person) but who have no suitably matched donors. The advantages of UCB are that (1) it is associated with less risk of transmitting an infection from a donor, (2) it can be more safely given even if not completely matched compared to bone marrow or blood stem cells, and (3) it is much more quickly available than unrelated donor bone marrow or blood stem cells. While more commonly used for transplantation in children, UCB is increasingly being used in adults. However, because they are larger than children, the relatively smaller stem cell dose in UCB is major limitation for transplantation in adults, and engraftment can be delayed. This study is investigating whether the drug sitagliptin can be used to increase and speed up engraftment in adults receiving UCB transplantation, overcoming the limitation of small stem cell doses associated with umbilical cord blood.

Sitagliptin is a drug given in tablet form that has been recently approved by the Food and Drug Administration (FDA) for the treatment of certain patients with diabetes mellitus (a disease that results in high blood sugar). Sitagliptin has been given to both normal healthy volunteers and diabetic patients and has been found to be safe and well-tolerated. The drug improves control of blood sugar in diabetics by inhibiting an enzyme called "CD26/DPP-IV." Recent studies at Indiana University (and other centers) have shown that this same enzyme plays an important role in the way transplanted stem cells find their way to the bone marrow and engraft. Transplant studies in mice have found that inhibiting CD26/DPP-IV significantly increases the engraftment of stem cells. Based on these studies, it is believed that drugs that inhibit CD26/DPP-IV, such as sitagliptin, may also increase engraftment in patients who receive clinical stem cell transplants.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following disease types with disease-specific features as outlined in the protocol:

  * Acute myeloid leukemia (AML)
  * Acute lymphoblastic leukemia (ALL)
  * Myelodysplasia
  * Chronic myelogenous leukemia
  * Patients with aggressive non-Hodgkin's lymphoma (NHL), including diffuse large cell lymphoma, mediastinal B-cell lymphoma, transformed lymphoma, mantle cell lymphoma, and peripheral T cell lymphoma
  * Hodgkin's lymphoma
  * Relapsed Multiple Myeloma
* At least 35 days following start of preceding leukemia induction cytotoxic chemotherapy
* Patient age 18-55 years
* Karnofsky Performance status ≥ 70%
* No availability of a consenting HLA-matched related donor who is either matched fully matched or mismatched at only one locus of HLA-A, -B, and DRB1.
* No availability of a readily available HLA-matched volunteer unrelated donor (8 of 8 allele match at HLA-A, -B, -C and -DRB1). Patients with unstable disease who are in danger of significant disease progression while waiting to procure volunteer donor cells will be eligible to be treated on this protocol, even if a matched donor is available.
* Patients must have a matched or partially matched UCB unit with greater than 1.8 x10-7 nucleated cells/kg of recipient weight at the time of cryopreservation.
* No current uncontrolled bacterial, viral or fungal infection (defined as currently taking medication and progression of clinical symptoms).
* No HIV disease. Patients with immune dysfunction are at a significantly higher risk of infection from intensive immunosuppressive therapies.
* Non pregnant and non-nursing. Treatment under this protocol would expose a fetus to significant risks.
* Required baseline laboratory values as defined in the protocol

Exclusion Criteria:

* Symptomatic uncontrolled coronary artery disease or congestive heart failure.
* Severe hypoxemia with room air PaO2 less than 70, supplemental oxygen dependence, or DLCO less than 50 percent predicted
* Patients with central nervous system (CNS) involvement refractory to intrathecal chemotherapy
* Prior allogeneic or autologous hematopoietic stem cell transplant in the last 6 months

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2009-03; Primary Completion 2012-11 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Farag, MD, PhD, Principal Investigator — IU Simon Cancer Center
Locations (1):
- IU Simon Cancer Center, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Farag SS, Srivastava S, Messina-Graham S, Schwartz J, Robertson MJ, Abonour R, Cornetta K, Wood L, Secrest A, Strother RM, Jones DR, Broxmeyer HE. In vivo DPP-4 inhibition to enhance engraftment of single-unit cord blood transplants in adults with hematological malignancies. Stem Cells Dev. 2013 Apr 1;22(7):1007-15. doi: 10.1089/scd.2012.0636. Epub 2013 Feb 15. PMID 23270493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initially based on single arm 2 stage design using 600 mg sitagliptin/24 hrs in RBC replete and RBC depleted UCB units. In an unplanned interim analysis after 1st 20 enrolled pts, protocol was amended to exclude RBC replete UCB units due to worse outcomes and to test more frequent dosing of sitagliptin due to suboptimal inhibition of plasma DPP-IV.
Groups:
- Red Cell-Depleted (RCD) - 600 mg Sitagliptin/24 Hrs: 600 mg sitagliptin/day PO starting on Day -1 for a total of 4 doses in red cell-depleted patients
- Red Cell-Replete, Plasma-Depleted (PD) - 600 mg Sitagliptin/24: 600 mg sitagliptin/day PO starting on Day -1 for a total of 4 doses in red cell-replete patients
- 600 mg Sitagliptin/12 Hrs: 600 mg sitagliptin/bid PO starting on Day -1 for a total of 8 doses
- 600 mg Sitagliptin/8 Hrs: 600 mg sitagliptin/tid PO starting on Day -1 for a total of 12 doses
Period: Overall Study
Arm/Group | Red Cell-Depleted (RCD) - 600 mg Sitagliptin/24 Hrs | Red Cell-Replete, Plasma-Depleted (PD) - 600 mg Sitagliptin/24 | 600 mg Sitagliptin/12 Hrs | 600 mg Sitagliptin/8 Hrs
Started | 17 | 7 | 4 | 1
Completed | 7 | 1 | 0 | 0
Not Completed | 10 | 6 | 4 | 1
Not completed — Disease Progression | 5 | 0 | 1 | 0
Not completed — Death | 5 | 6 | 1 | 1
Not completed — Engraftment failure | 0 | 0 | 1 | 0
Not completed — Veno-Occlusive Disease | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Red Cell-Depleted (RCD) - 600 mg Sitagliptin/24 Hrs | Red Cell-Replete, Plasma-Depleted (PD) - 600 mg Sitagliptin/24 | 600 mg Sitagliptin/12 Hrs | 600 mg Sitagliptin/8 Hrs | Total
Number analyzed (Participants) | 17 | 7 | 4 | 1 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 7 | 4 | 1 | 29
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (10.86) | 34.8 (8.95) | 46.9 (7.94) | 54.9 (0) | 40.6 (10.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 2 | 1 | 19
  Male | 5 | 3 | 2 | 0 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 7 | 4 | 1 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 0 | 0 | 5
  White | 14 | 5 | 4 | 1 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Patients With Engraftment by Day +30 Following Transplant
Description: Evaluate the efficacy of CD26/DPP-IV inhibition in increasing the cumulative incidence of adult patients with hematological malignancies engrafting by day +30 following transplantation of UCB by 30 percent. The cumulative incidence of patients achieving this will be reported. The value of the estimate will be from bootstrapping 1000 samples with replacement of the data and the 95% confidence interval will be calculated using the percentile method.
Time Frame: Transplant (Day 0) through Day +30
Population: Modified Intent to treat population (mITT) - all patients receiving at least one dose of study drug and receiving REB depleted UCB units only
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Red Cell-Depleted (RCD) - 600 mg Sitagliptin/24 Hrs
Number analyzed (Participants) | 17
percentage of participants | 88 [74 to 100]

2. Secondary Outcome: Time to Neutrophil Engraftment
Description: Time to neutrophil engraftment will be analyzed by the Kaplan-Meier method. The time to engraftment of neutrophils is defined as the time from day 0 to the date of the first of three consecutive days after transplantation during which the absolute neutrophils count (ANC) is at least 0.5 x109/l. Patients who did not have neutrophil engraftment before death will be censored at the date of death. The median and 95% confidence intervals will be provided. For the RCD group, all patients engrafted before day +30, except one patient who died at day 28 before engraftment. For the PD group, all patients engrafted before day +100, except one patient who died on day +103 before engraftment. For the 600 mg sitagliptin/12 hours group, two patients engrafted before day +100, and the other two patients died before day +100 before engraftment. The one patient on 600 mg sitagliptin/8 hours died on day +14 before engraftment.
Time Frame: Transplant (Day 0) up to 1 year
Population: All patients enrolled and received treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Red Cell-Depleted (RCD) - 600 mg Sitagliptin/24 Hrs | Red Cell-Replete, Plasma-Depleted (PD) - 600 mg Sitagliptin/24 | 600 mg Sitagliptin/12 Hrs | 600 mg Sitagliptin/8 Hrs
Number analyzed (Participants) | 17 | 7 | 4 | 1
days | 21 [15 to 25] | 35 [25 to 98] | 51 [23 to 95] | 14 [NA to NA] — Only 1 patient was in this group and so a 95% Confidence Interval was not able to be calculated.

3. Secondary Outcome: Time to Platelet Engraftment
Description: Time to platelet engraftment will be analyzed by the Kaplan-Meier method. The time to engraftment of platelets is defined as the time from day 0 to the first of seven consecutive days after transplantation during which the platelet count is at least 20 x109/l without transfusion support. Only patients who achieved engraftment of platelets will be included in the analysis. The median and 95% confidence intervals will be provided.
Time Frame: Transplant (Day 0) up to 1 year
Population: All patients enrolled and received treatment who achieved platelet recovery/engraftment of platelets.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Red Cell-Depleted (RCD) - 600 mg Sitagliptin/24 Hrs | Red Cell-Replete, Plasma-Depleted (PD) - 600 mg Sitagliptin/24 | 600 mg Sitagliptin/12 Hrs | 600 mg Sitagliptin/8 Hrs
Number analyzed (Participants) | 17 | 7 | 4 | 1
days | 77 [51 to 97] | 91 [80 to 102] | NA [NA to NA] — With few patients, the median was not able to be achieved and the 95% confidence interval could not be calculated. | NA [NA to NA] — With few patients, the median was not able to be achieved and the 95% confidence interval could not be calculated.

4. Secondary Outcome: Treatment Related Adverse Events Grade 3 or Higher for Non-hematological Toxicity
Description: Number of unique patients who had a treatment related (possible, probable or definite) non-hematological adverse event that was graded 3 or greater.
Time Frame: Transplant (Day 0) up to 3 years
Population: All patients enrolled and received treatment.
Measure: Number; unit: participants
Arm/Group | Red Cell-Depleted (RCD) - 600 mg Sitagliptin/24 Hrs | Red Cell-Replete, Plasma-Depleted (PD) - 600 mg Sitagliptin/24 | 600 mg Sitagliptin/12 Hrs | 600 mg Sitagliptin/8 Hrs
Number analyzed (Participants) | 17 | 7 | 4 | 1
participants | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: up to 3 years
Arm/Group | Red Cell-Depleted (RCD) - 600 mg Sitagliptin/24 Hrs | Red Cell-Replete, Plasma-Depleted (PD) - 600 mg Sitagliptin/24 | 600 mg Sitagliptin/12 Hrs | 600 mg Sitagliptin/8 Hrs
Serious Adverse Events (participants affected / at risk) | 11/17 | 6/7 | 2/4 | 1/1
Other Adverse Events (participants affected / at risk) | 17/17 | 7/7 | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Red Cell-Depleted (RCD) - 600 mg Sitagliptin/24 Hrs (N=17) | Red Cell-Replete, Plasma-Depleted (PD) - 600 mg Sitagliptin/24 (N=7) | 600 mg Sitagliptin/12 Hrs (N=4) | 600 mg Sitagliptin/8 Hrs (N=1)
BLOOD/BONE MARROW - OTHER (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
LYMPHATICS - OTHER (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
CARDIAC ARRHYTHMIA - OTHER (Cardiac disorders) | 1 | 0 | 0 | 0
CARDIAC GENERAL - OTHER (Cardiac disorders) | 0 | 0 | 0 | 1
RESTRICTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 | 1 | 0 | 0
DIARRHEA (Gastrointestinal disorders) | 4 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 3 | 0 | 0 | 0
PAIN - ABDOMEN NOS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 3 | 1 | 0 | 0
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 1 | 0 | 0 | 0
HYPOTHERMIA (General disorders) | 1 | 0 | 0 | 0
HEPATOBILIARY/PANCREAS - OTHER (Hepatobiliary disorders) | 0 | 0 | 1 | 0
LIVER DYSFUNCTION/FAILURE (CLINICAL) (Hepatobiliary disorders) | 0 | 1 | 0 | 0
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 1 | 0 | 0 | 0
FEBRILE NEUTROPENIA (FEVER OF UNKNOWN ORIGIN WITHOUT CLINICALLY OR MICROBIOLOGICALLY DOCUMENTED INFE (Infections and infestations) | 2 | 1 | 0 | 1
INFECTION (DOCUMENTED CLINICALLY OR MICROBIOLOGICALLY) WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E (Infections and infestations) | 4 | 1 | 0 | 0
INFECTION - OTHER (Infections and infestations) | 4 | 1 | 0 | 0
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - BLOOD (Infections and infestations) | 0 | 1 | 0 | 0
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - BRONCHUS (Infections and infestations) | 1 | 0 | 0 | 0
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - SINUS (Infections and infestations) | 1 | 0 | 0 | 0
INFECTION WITH UNKNOWN ANC - LUNG (PNEUMONIA) (Infections and infestations) | 1 | 1 | 0 | 0
INFECTION WITH UNKNOWN ANC - SINUS (Infections and infestations) | 1 | 0 | 0 | 0
CERVICAL SPINE-RANGE OF MOTION (Investigations) | 1 | 0 | 0 | 0
PAIN - EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
CONFUSION (Nervous system disorders) | 1 | 0 | 0 | 0
PAIN - HEAD/HEADACHE (Nervous system disorders) | 1 | 0 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 1 | 0
ADULT RESPIRATORY DISTRESS SYNDROME (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
EDEMA, LARYNX (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 1
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
PULMONARY/UPPER RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
HEMORRHAGE, GI - ABDOMEN NOS (Vascular disorders) | 1 | 0 | 0 | 0
HEMORRHAGE, GI - LOWER GI NOS (Vascular disorders) | 1 | 0 | 0 | 0
HEMORRHAGE, GU - URINARY NOS (Vascular disorders) | 0 | 1 | 0 | 0
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY - LUNG (Vascular disorders) | 1 | 0 | 0 | 0
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY - RESPIRATORY TRACT NOS (Vascular disorders) | 1 | 0 | 0 | 0
HYPOTENSION (Vascular disorders) | 1 | 0 | 0 | 1
VASCULAR - OTHER (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Red Cell-Depleted (RCD) - 600 mg Sitagliptin/24 Hrs (N=17) | Red Cell-Replete, Plasma-Depleted (PD) - 600 mg Sitagliptin/24 (N=7) | 600 mg Sitagliptin/12 Hrs (N=4) | 600 mg Sitagliptin/8 Hrs (N=1)
BLOOD/BONE MARROW - OTHER (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
COAGULATION - OTHER (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
HEMOLYSIS (E.G., IMMUNE HEMOLYTIC ANEMIA, DRUG-RELATED HEMOLYSIS) (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0
LYMPHATICS - OTHER (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
CARDIAC ARRHYTHMIA - OTHER (Cardiac disorders) | 5 | 4 | 1 | 1
CARDIAC GENERAL - OTHER (Cardiac disorders) | 3 | 3 | 0 | 0
PERICARDIAL EFFUSION (NON-MALIGNANT) (Cardiac disorders) | 3 | 2 | 0 | 0
RESTRICTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 | 1 | 0 | 0
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA - ATRIAL TACHYCARDIA/PAROXYSMAL ATRIAL TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA - SINUS BRADYCARDIA (Cardiac disorders) | 2 | 0 | 0 | 0
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA - SINUS TACHYCARDIA (Cardiac disorders) | 7 | 2 | 0 | 0
VALVULAR HEART DISEASE (Cardiac disorders) | 1 | 0 | 0 | 0
VENTRICULAR ARRHYTHMIA - VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0
AUDITORY/EAR - OTHER (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
PAIN - MIDDLE EAR (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
THYROID FUNCTION, LOW (HYPOTHYROIDISM) (Endocrine disorders) | 1 | 0 | 0 | 0
DRY EYE SYNDROME (Eye disorders) | 1 | 0 | 0 | 0
OPHTHALMOPLEGIA/DIPLOPIA (DOUBLE VISION) (Eye disorders) | 1 | 0 | 0 | 0
PAIN - EYE (Eye disorders) | 1 | 0 | 0 | 0
RETINAL DETACHMENT (Eye disorders) | 1 | 0 | 0 | 0
VISION-BLURRED VISION (Eye disorders) | 3 | 1 | 0 | 0
VISION-FLASHING LIGHTS/FLOATERS (Eye disorders) | 1 | 1 | 0 | 0
WATERY EYE (EPIPHORA, TEARING) (Eye disorders) | 0 | 1 | 0 | 0
ASCITES (NON-MALIGNANT) (Gastrointestinal disorders) | 4 | 0 | 1 | 0
COLITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
COLITIS, INFECTIOUS (E.G., CLOSTRIDIUM DIFFICILE) (Gastrointestinal disorders) | 1 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 4 | 3 | 1 | 0
DIARRHEA (Gastrointestinal disorders) | 17 | 7 | 4 | 1
DISTENSION/BLOATING, ABDOMINAL (Gastrointestinal disorders) | 4 | 1 | 2 | 0
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 2 | 1 | 0 | 0
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 1 | 2 | 0 | 0
FLATULENCE (Gastrointestinal disorders) | 1 | 0 | 0 | 0
GASTRITIS (INCLUDING BILE REFLUX GASTRITIS) (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 3 | 0 | 1 | 0
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 1 | 0 | 1 | 0
HEMORRHOIDS (Gastrointestinal disorders) | 1 | 1 | 0 | 0
HICCOUGHS (HICCUPS, SINGULTUS) (Gastrointestinal disorders) | 1 | 0 | 0 | 0
INCONTINENCE, ANAL (Gastrointestinal disorders) | 0 | 1 | 0 | 0
MUCOSITIS/STOMATITIS (CLINICAL EXAM) - ESOPHAGUS (Gastrointestinal disorders) | 1 | 0 | 1 | 0
MUCOSITIS/STOMATITIS (CLINICAL EXAM) - ORAL CAVITY (Gastrointestinal disorders) | 15 | 7 | 3 | 1
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) - ORAL CAVITY (Gastrointestinal disorders) | 1 | 1 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 15 | 5 | 4 | 1
OBSTRUCTION, GI - STOMACH (Gastrointestinal disorders) | 1 | 0 | 0 | 0
OCULAR/VISUAL - OTHER (Gastrointestinal disorders) | 1 | 0 | 0 | 0
PAIN - ABDOMEN NOS (Gastrointestinal disorders) | 13 | 3 | 3 | 0
PAIN - ANUS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
PAIN - DENTAL/TEETH/PERIDONTAL (Gastrointestinal disorders) | 0 | 0 | 1 | 0
PAIN - RECTUM (Gastrointestinal disorders) | 2 | 0 | 0 | 0
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 1 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 14 | 6 | 4 | 0
EDEMA: HEAD AND NECK (General disorders) | 3 | 1 | 1 | 1
EDEMA: LIMB (General disorders) | 12 | 4 | 2 | 1
EDEMA: TRUNK/GENITAL (General disorders) | 5 | 0 | 1 | 0
EDEMA: VISCERA (General disorders) | 1 | 0 | 0 | 0
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 2 | 3 | 0 | 0
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 14 | 4 | 2 | 0
PAIN - BUTTOCK (General disorders) | 0 | 1 | 0 | 0
PAIN - CHEST WALL (General disorders) | 2 | 2 | 0 | 0
PAIN - CHEST/THORAX NOS (General disorders) | 2 | 0 | 0 | 0
PAIN - OTHER (General disorders) | 11 | 3 | 1 | 1
PAIN - PAIN NOS (General disorders) | 3 | 0 | 0 | 0
RIGORS/CHILLS (General disorders) | 0 | 1 | 0 | 0
SWEATING (DIAPHORESIS) (General disorders) | 0 | 1 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0
HEPATOBILIARY/PANCREAS - OTHER (Hepatobiliary disorders) | 2 | 0 | 0 | 0
LIVER DYSFUNCTION/FAILURE (CLINICAL) (Hepatobiliary disorders) | 1 | 1 | 0 | 0
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 1 | 0 | 0 | 0
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Immune system disorders) | 7 | 0 | 0 | 0
ALLERGY/IMMUNOLOGY - OTHER (Immune system disorders) | 0 | 1 | 0 | 0
SERUM SICKNESS (Immune system disorders) | 1 | 0 | 0 | 0
FEBRILE NEUTROPENIA (FEVER OF UNKNOWN ORIGIN WITHOUT CLINICALLY OR MICROBIOLOGICALLY DOCUMENTED INFE (Infections and infestations) | 13 | 5 | 3 | 1
INFECTION (DOCUMENTED CLINICALLY OR MICROBIOLOGICALLY) WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E (Infections and infestations) | 11 | 4 | 2 | 0
INFECTION - OTHER (Infections and infestations) | 11 | 4 | 3 | 1
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - ANAL/PERIANAL (Infections and infestations) | 1 | 0 | 0 | 0
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - BLADDER (URINARY) (Infections and infestations) | 2 | 0 | 0 | 0
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - BLOOD (Infections and infestations) | 2 | 0 | 0 | 0
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - COLON (Infections and infestations) | 1 | 0 | 0 | 0
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - LUNG (PNEUMONIA) (Infections and infestations) | 1 | 0 | 0 | 0
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - PARANASAL (Infections and infestations) | 1 | 0 | 0 | 0
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - SINUS (Infections and infestations) | 1 | 0 | 0 | 0
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - SMALL BOWEL NOS (Infections and infestations) | 1 | 0 | 0 | 0
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - URINARY TRACT NOS (Infections and infestations) | 3 | 0 | 0 | 0
INFECTION WITH UNKNOWN ANC - BLADDER (URINARY) (Infections and infestations) | 1 | 0 | 1 | 0
INFECTION WITH UNKNOWN ANC - BLOOD (Infections and infestations) | 0 | 1 | 0 | 0
INFECTION WITH UNKNOWN ANC - COLON (Infections and infestations) | 2 | 1 | 0 | 0
INFECTION WITH UNKNOWN ANC - CONJUNCTIVA (Infections and infestations) | 0 | 1 | 0 | 0
INFECTION WITH UNKNOWN ANC - EYE NOS (Infections and infestations) | 2 | 0 | 0 | 0
INFECTION WITH UNKNOWN ANC - LUNG (PNEUMONIA) (Infections and infestations) | 2 | 2 | 0 | 0
INFECTION WITH UNKNOWN ANC - MIDDLE EAR (OTITIS MEDIA) (Infections and infestations) | 1 | 0 | 0 | 0
INFECTION WITH UNKNOWN ANC - SINUS (Infections and infestations) | 6 | 1 | 0 | 0
INFECTION WITH UNKNOWN ANC - SKIN (CELLULITIS) (Infections and infestations) | 1 | 0 | 0 | 0
INFECTION WITH UNKNOWN ANC - SOFT TISSUE NOS (Infections and infestations) | 0 | 1 | 0 | 0
INFECTION WITH UNKNOWN ANC - UPPER AIRWAY NOS (Infections and infestations) | 3 | 1 | 0 | 0
INFECTION WITH UNKNOWN ANC - URINARY TRACT NOS (Infections and infestations) | 1 | 0 | 0 | 0
WOUND COMPLICATION, NON-INFECTIOUS (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
ALKALINE PHOSPHATASE (Investigations) | 15 | 4 | 2 | 0
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 17 | 4 | 3 | 1
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 17 | 6 | 4 | 1
BICARBONATE, SERUM-LOW (Investigations) | 2 | 0 | 0 | 0
CARDIAC TROPONIN I (CTNI) (Investigations) | 0 | 0 | 0 | 1
CREATININE (Investigations) | 12 | 5 | 3 | 1
HAPTOGLOBIN (Investigations) | 0 | 0 | 1 | 0
HEMOGLOBIN (Investigations) | 2 | 0 | 0 | 0
ILEUS, GI (FUNCTIONAL OBSTRUCTION OF BOWEL, I.E., NEUROCONSTIPATION) (Investigations) | 0 | 0 | 1 | 0
METABOLIC/LABORATORY - OTHER (Investigations) | 5 | 1 | 2 | 0
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Investigations) | 1 | 0 | 0 | 0
PLATELETS (Investigations) | 1 | 2 | 0 | 0
PROLONGED QTC INTERVAL (Investigations) | 0 | 1 | 0 | 0
WEIGHT GAIN (Investigations) | 2 | 0 | 2 | 0
WEIGHT LOSS (Investigations) | 1 | 0 | 0 | 0
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Metabolism and nutrition disorders) | 11 | 4 | 3 | 1
ANOREXIA (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
BILIRUBIN (HYPERBILIRUBINEMIA) (Metabolism and nutrition disorders) | 15 | 6 | 2 | 1
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Metabolism and nutrition disorders) | 8 | 3 | 3 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Metabolism and nutrition disorders) | 10 | 3 | 3 | 0
GLUCOSE, SERUM-LOW (HYPOGLYCEMIA) (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Metabolism and nutrition disorders) | 7 | 3 | 2 | 0
PHOSPHATE, SERUM-LOW (HYPOPHOSPHATEMIA) (Metabolism and nutrition disorders) | 7 | 4 | 3 | 0
POTASSIUM, SERUM-HIGH (HYPERKALEMIA) (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Metabolism and nutrition disorders) | 5 | 5 | 2 | 0
SODIUM, SERUM-HIGH (HYPERNATREMIA) (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0
SODIUM, SERUM-LOW (HYPONATREMIA) (Metabolism and nutrition disorders) | 6 | 1 | 0 | 0
TRIGLYCERIDE, SERUM-HIGH (HYPERTRIGLYCERIDEMIA) (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
FRACTURE (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) - EXTREMITY-LOWER (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) - EXTREMITY-UPPER (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) - WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
MUSCULOSKELETAL/SOFT TISSUE - OTHER (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
PAIN - BACK (Musculoskeletal and connective tissue disorders) | 8 | 1 | 1 | 0
PAIN - BONE (Musculoskeletal and connective tissue disorders) | 6 | 0 | 0 | 0
PAIN - EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1 | 0
PAIN - JOINT (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
PAIN - MUSCLE (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0
PAIN - NECK (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
SOFT TISSUE NECROSIS - EXTREMITY-LOWER (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
CONFUSION (Nervous system disorders) | 7 | 3 | 1 | 0
DIZZINESS (Nervous system disorders) | 5 | 0 | 0 | 1
ENCEPHALOPATHY (Nervous system disorders) | 3 | 2 | 2 | 0
EXTRAPYRAMIDAL/INVOLUNTARY MOVEMENT/RESTLESSNESS (Nervous system disorders) | 1 | 0 | 0 | 0
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 2 | 0 | 0
MOOD ALTERATION - AGITATION (Nervous system disorders) | 1 | 0 | 1 | 0
MOOD ALTERATION - ANXIETY (Nervous system disorders) | 2 | 1 | 0 | 0
MOOD ALTERATION - DEPRESSION (Nervous system disorders) | 4 | 1 | 0 | 0
NEUROLOGY - OTHER (Nervous system disorders) | 2 | 0 | 0 | 0
NEUROPATHY: MOTOR (Nervous system disorders) | 0 | 1 | 0 | 0
NEUROPATHY: SENSORY (Nervous system disorders) | 7 | 1 | 2 | 0
PAIN - HEAD/HEADACHE (Nervous system disorders) | 9 | 4 | 1 | 1
PAIN - NEURALGIA/PERIPHERAL NERVE (Nervous system disorders) | 0 | 1 | 0 | 0
SEIZURE (Nervous system disorders) | 1 | 1 | 0 | 0
SOMNOLENCE/DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 2 | 0
SYNCOPE (FAINTING) (Nervous system disorders) | 1 | 0 | 0 | 0
TREMOR (Nervous system disorders) | 4 | 4 | 0 | 0
INSOMNIA (Psychiatric disorders) | 3 | 3 | 0 | 0
PSYCHOSIS (HALLUCINATIONS/DELUSIONS) (Psychiatric disorders) | 0 | 1 | 0 | 0
BLADDER SPASMS (Renal and urinary disorders) | 6 | 2 | 1 | 0
CYSTITIS (Renal and urinary disorders) | 2 | 1 | 0 | 0
INCONTINENCE, URINARY (Renal and urinary disorders) | 0 | 1 | 0 | 0
PAIN - BLADDER (Renal and urinary disorders) | 2 | 1 | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0 | 2 | 1
RENAL/GENITOURINARY - OTHER (Renal and urinary disorders) | 1 | 1 | 0 | 1
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 2 | 1 | 0 | 0
URINE COLOR CHANGE (Renal and urinary disorders) | 0 | 1 | 0 | 0
IRREGULAR MENSES (CHANGE FROM BASELINE) (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
PAIN - PELVIS (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
PAIN - URETHRA (Reproductive system and breast disorders) | 2 | 0 | 1 | 0
PAIN - VAGINA (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
VAGINAL DISCHARGE (NON-INFECTIOUS) (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
VAGINAL DRYNESS (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
PAIN - THROAT/PHARYNX/LARYNX (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0
ADULT RESPIRATORY DISTRESS SYNDROME (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
BRONCHOSPASM, WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 0 | 1
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 3 | 0
EDEMA, LARYNX (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 11 | 4 | 1 | 1
NASAL CAVITY/PARANASAL SINUS REACTIONS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 1 | 1
PNEUMONITIS/PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
PULMONARY/UPPER RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 1
VOICE CHANGES/DYSARTHRIA (E.G., HOARSENESS, LOSS OR ALTERATION IN VOICE, LARYNGITIS) (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
DERMATOLOGY/SKIN - OTHER (Skin and subcutaneous tissue disorders) | 5 | 2 | 2 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
PAIN - SKIN (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 6 | 1 | 1 | 0
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 6 | 3 | 0 | 0
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 7 | 0 | 2 | 0
RASH: DERMATITIS ASSOCIATED WITH RADIATION - RADIATION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
RASH: ERYTHEMA MULTIFORME (E.G., STEVENS-JOHNSON SYNDROME, TOXIC EPIDERMAL NECROLYSIS) (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
RASH: HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
SKIN BREAKDOWN/DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
ULCERATION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
HEMORRHAGE, CNS (Vascular disorders) | 0 | 0 | 0 | 1
HEMORRHAGE, GI - ABDOMEN NOS (Vascular disorders) | 4 | 1 | 0 | 0
HEMORRHAGE, GI - ANUS (Vascular disorders) | 1 | 0 | 0 | 0
HEMORRHAGE, GI - LOWER GI NOS (Vascular disorders) | 2 | 1 | 1 | 0
HEMORRHAGE, GI - UPPER GI NOS (Vascular disorders) | 1 | 1 | 0 | 0
HEMORRHAGE, GU - BLADDER (Vascular disorders) | 4 | 1 | 0 | 0
HEMORRHAGE, GU - URINARY NOS (Vascular disorders) | 5 | 3 | 2 | 0
HEMORRHAGE, GU - VAGINA (Vascular disorders) | 4 | 2 | 0 | 0
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY - BRONCHOPULMONARY NOS (Vascular disorders) | 0 | 1 | 0 | 0
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY - NOSE (Vascular disorders) | 5 | 0 | 0 | 0
HEMORRHAGE/BLEEDING - OTHER (Vascular disorders) | 0 | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 6 | 2 | 0 | 0
HYPOTENSION (Vascular disorders) | 9 | 3 | 3 | 0
PERIPHERAL ARTERIAL ISCHEMIA (Vascular disorders) | 0 | 0 | 0 | 1
PULMONARY HYPERTENSION (Vascular disorders) | 1 | 0 | 0 | 0
VASCULAR - OTHER (Vascular disorders) | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes